CLINICAL TRIAL: NCT00471640
Title: Dexamethasone Infusion in Community-acquired Pneumonia
Acronym: Ovidius
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: St. Antonius Hospital (Other)
Responsible Party: St. Antonius Hospital, St. Antonius Hospital
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: versie 1
Record Dates: First submitted 2007-05-08; First posted 2007-05-10 (Estimated); Last update posted 2010-09-27 (Estimated); Status verified 2010-09

CONDITIONS: Pneumonia
Keywords: pneumonia; dexamethasone; community-acquired pneumonia
MeSH Terms: conditions — Pneumonia; Community-Acquired Pneumonia | interventions — Dexamethasone

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- 1 (Active Comparator): dexamethasone
  Interventions: Drug: dexamethasone
- 2 (Placebo Comparator): Placebo
  Interventions: Drug: dexamethasone

INTERVENTIONS:
Drug: dexamethasone — 4 days 5 mg

SUMMARY:
The purpose of this study is to determine whether dexamethasone reduces the length of hospital stay in patient with a community-acquired pneumonia.

DETAILED DESCRIPTION:
Community-acquired pneumonia (CAP) is common and approximately 20 percent of all episodes of pneumonia result in hospitalization. It is the leading cause of community-acquired infection requiring ICU admission.1 Especially elderly patients may have a severe illness with a high morbidity and mortality rate. In pulmonary infections, the release of cytokines and other inflammatory mediators from alveolar macrophages serves as a useful mechanism in the elimination of invading pathogens. However, this natural reaction can be potentially harmful when excessive release of circulating inflammatory cytokines causes damage to the patient, particularly the lung.

Interest in the role of corticosteroids in the pathophysiology of critical illness has existed since the early part of the 20th century. On ICU, early treatment with corticosteroids to attenuate systemic inflammation is widespread. At the same time, outside the ICU little evidence is available on the effect of treatment with corticosteroids in patients diagnosed with CAP. Hypothetically, early initiated administration of corticosteroids in the course of a CAP can lower systemic and pulmonary inflammation. This may lead to earlier resolution of pneumonia and a reduction of complications (sepsis, mortality).

ELIGIBILITY:
Inclusion Criteria:

Patients aged 18 to 100 years with a community-acquired pneumonia.

Criteria to determine a community-acquired pneumonia:

* Chest radiograph showing new opacities
* In combination with two of the following findings:

  * Cough
  * Production of sputum
  * Temp >38,0 °C or <36,0 °C
  * Audible abnormalities by chest examination compatible with pneumonia
  * Leukocytosis (>10.000 cells/mm3), leftward shift (>10%) or leukopenia (<4000 cells/mm3)
  * CRP > 15 mg/dl (three times upper limit of normal)

Exclusion Criteria:

* o The following groups are excluded:

  * Immunocompromised patients:

    * Patients with a known congenital or achieved immunodeficiency.
    * Patients who received chemotherapy less than 6 weeks ago.
    * Patients who received corticosteroids in the last 6 weeks.
    * Patients who received immunosuppressive medication in the last 6 weeks. (like cyclosporine, cyclofosfamide, azathioprine)
    * Patients with COPD who are on systemic corticosteroids for COPD.
    * Patients who require ICU treatment.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 300 (Estimated)
Dates: Start 2007-11; Primary Completion 2010-09 (Actual); Study Completion 2010-09 (Actual)

PRIMARY OUTCOMES:
length of hospital stay | 30 days

SECONDARY OUTCOMES:
side-effects inflammation markers lung function | 30 days

CONTACTS AND LOCATIONS:
Overall Officials: D Biesma, dr., Study Director — St. Antonius Hospital
Locations (2):
- Netherlands (2):
  - Gelderse Vallei Ede, Ede, Gelderland
  - St Antonius Hosptial, Nieuwegein, Utrecht

REFERENCES:
- [Derived] Raeven VM, Spoorenberg SM, Boersma WG, van de Garde EM, Cannegieter SC, Voorn GP, Bos WJ, van Steenbergen JE; Alkmaar study group; Ovidius study group. Atypical aetiology in patients hospitalised with community-acquired pneumonia is associated with age, gender and season; a data-analysis on four Dutch cohorts. BMC Infect Dis. 2016 Jun 17;16:299. doi: 10.1186/s12879-016-1641-9. PMID 27317257
- [Derived] Remmelts HH, van de Garde EM, Meijvis SC, Peelen EL, Damoiseaux JG, Grutters JC, Biesma DH, Bos WJ, Rijkers GT. Addition of vitamin D status to prognostic scores improves the prediction of outcome in community-acquired pneumonia. Clin Infect Dis. 2012 Dec;55(11):1488-94. doi: 10.1093/cid/cis751. Epub 2012 Aug 31. PMID 22942205
- [Derived] Meijvis SC, Hardeman H, Remmelts HH, Heijligenberg R, Rijkers GT, van Velzen-Blad H, Voorn GP, van de Garde EM, Endeman H, Grutters JC, Bos WJ, Biesma DH. Dexamethasone and length of hospital stay in patients with community-acquired pneumonia: a randomised, double-blind, placebo-controlled trial. Lancet. 2011 Jun 11;377(9782):2023-30. doi: 10.1016/S0140-6736(11)60607-7. Epub 2011 Jun 1. PMID 21636122